CLINICAL TRIAL: NCT06761391
Title: Immediate Effects of Suboccipital Myofascial Release on Pain Pressure Threshold, Range of Motion, Balance, and Proprioception
Brief Title: Effects of Suboccipital Release on Sensorial and Functional Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bvu1903
Record Dates: First submitted 2024-12-22; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Suboccipital Muscles
Keywords: suboccipital release; neck proprioception; pain pressure threshold

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital Myofascial Release (Experimental): The application will be done in the supine position. The therapist will sit on the stool at the head of the stretcher with his/her forearm in contact with the stretcher. After palpating the occiput condyles with his/her fingers, the therapist will place his/her fingers in the slightly concave area between the occiput and the spinous process of the second cervical vertebra. The therapist will lift the participant's head a little by bending the metacarpophalangeal joints. While the base of the participant's skull is in the therapist's palm, the therapist will apply pressure equal to the weight of the participant's head with his/her second, third and fourth fingers on the participant's rectus capitis posterior and obliqus capitis superior muscles for 5 minutes. In order for eye movements not to affect the suboccipital muscle tone, the participants will be asked to close their eyes during the application.
  Interventions: Diagnostic Test: Pain Pressure Threshold; Diagnostic Test: Cervical Range of Motion; Diagnostic Test: Balance Error Scoring; Diagnostic Test: Cervical Joint Position Sense; Other: Suboccipital manual therapy
- Suboccipital Hold (Sham Comparator): No suboccipital relaxation will be applied to the control group, and the experimental group will be kept in contact with the suboccipital region for the same period of time, namely 5 minutes, and the measurements will be recorded before and after the application.
  Interventions: Diagnostic Test: Pain Pressure Threshold; Diagnostic Test: Cervical Range of Motion; Diagnostic Test: Balance Error Scoring; Diagnostic Test: Cervical Joint Position Sense; Other: Suboccipital manual therapy

INTERVENTIONS:
Diagnostic Test: Pain Pressure Threshold — A hand-held pressure algometer will be used to record the pressure pain threshold (PPT), defined as the level at which gradually increasing pressure becomes painful. Pressure algometry has shown high intratest reliability in asymptomatic individuals over the suboccipital area and upper trapezius. PPT levels will be measured bilaterally over the neck angle over the middle of the anterior surface of the upper trapezius; and over the rectus capitis posterior major (RCPM) muscle. The physiotherapist will use an increasing pressure of approximately 1 kg/cm²/s. The average of three measurements with a 30-second rest period will be taken for analysis. Two measurements will be taken, before and after.
Diagnostic Test: Cervical Range of Motion — The degrees obtained as a result of the Range of Motion (ROM) measurements are made with a universal manual goniometer. Goniometer is still the most commonly used method for ROM measurements. For all ROM measurements to be performed, the necessary measurements can be taken based on the American Academy of Orthopaedic Surgeons (AAOS) guidelines . The flexion, extension, right and left rotation angles of the cervical region will be measured and recorded with the goniometer in the sitting position of the person. The measurement will be made twice, before and after the application.
Diagnostic Test: Balance Error Scoring — Balance performance will be assessed using the Balance Error Scoring System (BESS), known in Turkish as DHPS. Subjects must maintain test positions for 20 seconds under 6 conditions with eyes closed and no support: 2 surfaces (flat and foam) and 3 stance positions (double-foot, single-foot, tandem). A laboratory floor will serve as the flat surface, and an exercise mat will serve as the foam surface. All subjects will perform the conditions in this sequence: double-foot flat, single-foot flat, tandem flat, double-foot foam, single-foot foam, tandem foam, both pre-test and post-test. Each 20-second period will be timed with a stopwatch, and each error within this period will count as 1 point. Each test condition has a maximum error score of 10. Errors include:
  1. Lifting hands above the iliac crest,
  2. Opening eyes,
  3. Taking a step,staggering, falling,
  4. Flexing or abducting the hip joint beyond 30°,
  5. Lifting the forefoot or heel off the ground,
  6. Leaving the test position
Diagnostic Test: Cervical Joint Position Sense — The sense of joint position in the cervical region will be evaluated in four positions: flexion, extension, right rotation, and left rotation, using a goniometer. Participants will sit upright with arms at their sides, looking ahead. The physiotherapist will passively move the participant's head to 65% of the maximum joint range of motion, previously determined, minimizing vestibular function effects. After holding the head in position for three seconds, participants will be asked to remember the position. Subsequently, they will be instructed to return their head to the neutral position and then actively move it to the previously determined point. The degree of error between the target and achieved positions will be measured.
Other: Suboccipital manual therapy — The procedure will be conducted with the patient lying on their back. The practitioner will be seated on a stool at the top of the examination table, their forearm in contact with the surface. After locating the occipital condyles through palpation, the practitioner will position their fingers in the slightly concave region between the occiput and the second cervical vertebra's spinous process. The patient's head will be gently elevated by the practitioner flexing their metacarpophalangeal joints. With the patient's skull base resting in the practitioner's palm, pressure equivalent to the weight of the patient's head will be applied to the rectus capitis posterior and obliquus capitis superior muscles using the practitioner's second, third, and fourth fingers for a duration of 5 minutes. To prevent eye movements from influencing suboccipital muscle tone, patients will be instructed to keep their eyes closed during the procedure.

SUMMARY:
Suboccipital release is a straightforward technique beneficial for addressing musculoskeletal complaints like neck pain and headaches. This versatile method aids the autonomic system by manipulating the occipital-atlanto region, specifically regulating the parasympathetic system rather than the sympathetic system targeted by most osteopathic treatments. Studies indicate this technique enhances range of motion and balance in the lower extremities of both healthy and pre-existing patients due to fascia connections throughout the body. Suboccipital muscle release increases cervical spine range of motion, facilitating physical therapy. Myofascial release significantly boosts joint flexibility and range of motion (ROM) without reducing strength or performance. The rectus capitus posterior minor (RCPM) muscle, dense with spindles, is crucial in the suboccipital region for balance and pain proprioception. Trauma-induced atrophy in this muscle is strongly linked to chronic neck pain and reduced standing balance. A case report showed that a patient undergoing a personalized balance program exhibited significant balance improvement, suggesting that balance training should be considered for cervicogenic pain intervention strategies. Neck muscle spasms or fatigue can impair proprioception and postural control, with prolonged unilateral cervical muscle contraction increasing neck proprioceptor sensitivity. Muscle fatigue-related interstitial inflammatory mediators can sensitize muscle spindles. This study will explore suboccipital relaxation's acute effects on pressure pain threshold, range of motion, balance, and joint position sense in healthy individuals based on existing literature.

DETAILED DESCRIPTION:
Suboccipital release is a relatively easy technique that a person can use to help with musculoskeletal complaints such as neck pain and headaches. This technique is also very versatile and can help regulate the autonomic system in the body due to the manipulation of the occipital-atlanto region. This technique has been noted to regulate the parasympathetic system rather than the sympathetic system that most osteopathic treatments target. Studies have shown that this technique improves range of motion and balance in the lower extremities of healthy and pre-existing patients due to the connection of the fascia throughout the body. The release of the suboccipital muscles increases the range of motion of the cervical spine, which makes it easier for the physical therapist. Myofascial release has been shown to significantly increase joint flexibility and range of motion (ROM) without causing any loss of strength or decreased performance . Studies on the rectus capitus posterior minor (RCPM) muscle indicate that it is one of the most important muscles in the suboccipital region. Because of the high density of muscle spindles, it is presumed that this muscle plays a role as a proprioceptive monitor important for balance and pain. Trauma has been shown to cause atrophy in this muscle, and this atrophy is strongly associated with chronic neck pain and decreased standing balance (4). A case report has shown that a patient who underwent a personalized balance program showed significant improvement in balance as measured by sensory organization testing; this improved balance control suggests that balance training should be considered when determining appropriate intervention strategies for patients with cervicogenic pain. Neck muscle spasms or fatigue can alter proprioception and postural control, and prolonged contraction of unilateral cervical muscles can significantly increase the sensitivity of neck proprioceptors. Interstitial inflammatory mediators produced by muscle fatigue can sensitize muscle spindles. The acute effects of suboccipital relaxation on pressure pain threshold, range of motion, balance, and joint position sense in healthy individuals have been examined in the literature.

ELIGIBILITY:
Inclusion Criteria:

Volunteers willing to participate in the study.

Exclusion Criteria:

Diagnosed with an upper extremity musculoskeletal system disease. Experiencing chronic headaches or migraine complaints. Presence of any pathology causing sensory or balance impairments. Diagnosed with a pathology in the cervical regio

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-02 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Neck Proprioception | Change from baseline to final examination immediate after 5 minutes of manual therapy
  Cervical Joint Position Sense Assessment was performed with the Reposition Test using a goniometer.

SECONDARY OUTCOMES:
Pain Pressure Threshold | Change from baseline to final examination immediate after 5 minutes of manual therapy
  Pain pressure threshold of the upper trapezius and rectus capitis muscles was measured with a handheld algometer
Range of Motion | Change from baseline to final examination immediate after 5 minutes of manual therapy
  A goniometer was utilized to assess the range of motion for cervical flexion, extension, and rotation.
Balance Error Scoring | Change from baseline to final examination immediate after 5 minutes of manual therapy
  Balance Error Scoring System was used to measure balance performances.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Safran E, Kaya Y. Contextual and placebo effects of suboccipital myofascial release: evaluating its influence on pain threshold, cervical range of motion, and proprioception. BMC Musculoskelet Disord. 2025 May 21;26(1):502. doi: 10.1186/s12891-025-08741-6. PMID 40399920